CLINICAL TRIAL: NCT06222736
Title: Evaluation of the Efficacy of Cervical Core Exercises in Persons With Temporomandibular Joint Dysfunction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Gelisim University (Other)
Responsible Party: Principal Investigator, Tuğçe Bilgiç, Lecturer, Istanbul Gelisim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IstanbulGelisimU
Record Dates: First submitted 2024-01-09; First posted 2024-01-25 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Temporomandibular Joint Disorders
Keywords: Temporomandibular Joint; servical core exercise; myofasial pain
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Intervention Model Description: Our study will be conducted at the Istanbul University-Çapa Faculty of Dentistry Total and Partial Prosthesis clinic with volunteers who have been diagnosed with Temporomandibular disfunction.
Who Masked: Participant
Masking Description: The numbers determined using the Research Randomiser program will be placed in an opaque envelope, and participants will be asked to choose an envelope. Participants will be included in groups according to the number they choose.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rocabado exercises group (Experimental): The most commonly known form of exercise for Temporomandibular Disfunction is Rocabado exercises, which use 6 types of exercises 6 times a day.
  Interventions: Other: Rocabado Exercises
- Servical Core Exercises Group (Experimental): The purpose of core exercises is to support the vertebral column, especially by activating the stabilizing muscles, and to develop and maintain proper cervical posture by increasing kinesthetic awareness. At the beginning of the exercises, the patient is taught to contract the deep stabilizer muscles in a controlled manner, in isolation, without contraction of the superficial muscles. Exercises 2 days a week for 8 weeks, maximum 30 minutes. The session will be actively applied by the patient for a period of time.
  Interventions: Other: Servical Core Exercises
- Rocabado Exercises and Servical Core Exercises Group (Experimental): The most commonly known form of exercise for Temporomandibular Disfunction is Rocabado exercises, which use 6 types of exercises 6 times a day. The purpose of Servical Core exercises is to support the vertebral column, especially by activating the stabilizing muscles, and to develop and maintain proper cervical posture by increasing kinesthetic awareness. At the beginning of the exercises, the patient is taught to contract the deep stabilizer muscles in a controlled manner, in isolation, without contraction of the superficial muscles. Exercises 2 days a week for 8 weeks, maximum 30 minutes. The session will be actively applied by the patient for a period of time.
  Interventions: Other: Rocabado Exercises; Other: Servical Core Exercises

INTERVENTIONS:
Other: Rocabado Exercises — Patients trained by Rocabado Exercises
  Arms: Rocabado Exercises and Servical Core Exercises Group; Rocabado exercises group
Other: Servical Core Exercises — Servical Core Exercises
  Arms: Rocabado Exercises and Servical Core Exercises Group; Servical Core Exercises Group

SUMMARY:
The aim is to reveal to what extent cervical core exercises affect the results of treatment in patients with Temporomandibular Joint Dysfunction caused by Myofascial pain syndrome. Randomization will be carried out by dividing individuals who agree to participate in the study into 3 groups of 20 people.Participants will be divided into three groups, and all three groups will receive treatment in 30-45 minute sessions a day, 2 days a week for 8 weeks.

DETAILED DESCRIPTION:
The aim is to reveal to what extent cervical core exercises affect the results of treatment in patients with Temporomandibular Joint Dysfunction caused by Myofascial pain syndrome. Randomization will be carried out by dividing individuals who agree to participate in the study into 3 groups of 20 people with the "Research Randomizer" program. Randomization, evaluation and treatment of the groups will be done by different researchers.

Participants will be divided into three groups, and all three groups will receive treatment in 30-45 minute sessions a day, 2 days a week for 8 weeks. Evaluation will be made at the beginning and at the eight week to see the short-term effects. Rocabado exercises will be given to the first group, Cervical Core exercises will be given to the second group, and Rocabado and Cervical Core exercises will be given together to the third group. After the initial evaluations, all exercises will be taught to the patients in the first week, they will be planned as home exercises in the following weeks, and online follow-up will be done via tele-rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with Temporomandibular Disorder caused by Myofascial Pain Syndrome
* Female gender aged 18 and over
* Volunteering to participate in the study
* Not having communication difficulties such as speaking and understanding Turkish or not being able to understand the exercises.

Exclusion Criteria:

* Having a history of acute trauma in and around the Temporomandibular Joint
* Having Temporomandibular Joint dysfunction due to neurological disease
* Having a history of surgical/invasive procedures or treatments on the Temporomandibular Joint
* Presence of infection or tumoral structure within intraoral structures
* Having a history of tooth loss or prosthetic tooth use
* Having a history of surgical procedure in the cervical area

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Temporomandibular disorders are limited to one gender due to the large female population.
Enrollment: 60 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-11-15 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | 8 weeks
  The severity of pain felt by individuals in the Temporomandibular Joint and Cervical Region, at rest, during activity and at night, will be evaluated numerically using the visual analog scale. Individuals will be told that the number "0" on a 10 cm horizontal line indicates "no pain" and the number "10" indicates "unbearable pain". The location marked by the individual will be determined as the pain intensity in cm.
Algometer | 8 weeks
  Algometer will be used for objective measurement of Pain Threshold Assessment. The pressure will be applied to the massater, temporalis and upper trapezius muscles bilaterally, increasing the pressure by 1kg/cm2 every three seconds until the patient feels pain. The subject is told to report when he/she feels pain while applying force (kg/cm²) with the device. This process is repeated three times to calculate the average value on the muscles.
Mandibular Range of Motion | 8 weeks
  Mandibular Range of Motion, Pain-free mouth opening, maximum mouth opening, maximum assisted mouth opening, right lateral and left lateral movements will be evaluated by the physiotherapist with the help of a ruler
Jaw Functionality Assessment | 8 weeks
  'Functional Limitation Scale of the Jaw-8' will be used for functionality evaluation. The individual is asked to determine the level of restriction for each of the 8 items on the scale in the last month. Individuals are told that the number '0' on a 10cm horizontal line indicates 'no restriction' and the number '10' indicates 'severe restriction'. Functionality limitation is calculated by taking the average of the individual's answers.
craniovertebral angle | 8 weeks
  An objective method of assessing cervical anterior tilt is to measure the craniovertebral angle. Head position is expressed in degrees (°) by measuring the angle between the horizontal plane and the seventh cervical vertebra (C7) and the ear with a goniometer. Measurements are taken while individuals sit in a comfortable position with their arms at their sides and their backs supported on a chair. C7 is detected by manual palpation. While one of the goniometric arms extends to the ear (external auditory canal), the other arm is kept parallel to the horizontal plane. C7, the angle between the ear and the horizontal plane is recorded in degrees
Cervical Range of Motion | 8 weeks
  The cervical region will be evaluated with the active Cervical Range of Motion device. The device consists of inclinometers placed on the left lateral side of the head, in the middle of the forehead and on the head, and a magnetic collar placed on the neck. All measurements will be made while patients are sitting in an upright position on a chair with their arms adjacent to the body.
Cervical region deep flexor muscle endurance | 8 weeks
  To evaluate deep flexor muscle endurance in the cervical region, the patient is placed on the abdomen with hands free while the patient is in a supine hook position. Isometrically lifts the patient's head 2.5 cm off the ground with the patient's chin at maximum tilt. The maximum time in which the patient raises his head and maintains this position is recorded in seconds. The test is terminated when the patient feels pain and cannot maintain the position.

SECONDARY OUTCOMES:
Neck Disability Assessment | 8 weeks
  The Neck Disability Index is a tool used to determine how the pain participants feel in their neck affects their daily lives. In the 10-question survey, A = 0 points, B = 1 point, C = 2 points, D = 3 points, E = 4 points, F = 5 points are given for each question and the total score is obtained. According to the test scoring, 0-4=No disability, 5-14=Mild disability, 15-24=Moderate disability, 25-34=Severe disability, 35 or above=Complete disability.
Psychiatric Evaluation | 8 weeks
  Hospital Anxiety and Depression Scale is used to determine individuals' depression and anxiety levels. The scale consists of two subscales, seven measuring anxiety and seven measuring depression (odd numbers are anxiety, even numbers are depression), and a total of 14 items. Each item is scored on a 4-point Likert scale between 0 and 3. According to the scores obtained from the scales, the anxiety and depression status of individuals is evaluated as not being sick (0-7 points), borderline sick (8-10 points), and significantly sick (11-21). Considering the cut-off scores in Turkey, which are affected by the cultural situation in the country, individuals who score 10 points or more from the anxiety subscale and individuals who score above 7 points from the depression subscale are defined as risky.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Gelisim University, Istanbul, Avcılar, Turkey (Türkiye)